CLINICAL TRIAL: NCT01913639
Title: Phase II Study of FOLFOX Plus Regorafenib in Patients With Unresectable or Metastatic Esophagogastric Cancer
Brief Title: FOLFOX Plus Regorafenib in Patients With Unresectable or Metastatic Esophagogastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-080
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: BAY 73-4506 (REGORAFENIB); FLUOROURACIL; LEUCOVORIN; OXALIPLATIN
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — regorafenib; Fluorouracil; Leucovorin; Oxaliplatin

ARMS (1):
- FOLFOX Plus Regorafenib (Experimental): Regorafenib 160 mg daily on days 4 to 10 and days 18 to 24 as four 40 mg coprecipitate tablets + mFOLFOX on Day 1 and Day 15 of each cycle. Each cycle consists of 28 days. All patients will receive systemic chemotherapy with the mFOLFOX regimen and regorafenib. The specific version of the FOLFOX regimen used at MSKCC is mFOLFOX6. mFOLFOX6 will be given on Day 1 of each cycle. Patients will receive Oxaliplatin 85 mg/m2 IV (over 120 minutes), leucovorin 400 mg/m2 IV (over 120 minutes), 5-FU 400 mg/m2 IVP, and 5-FU 1200 mg/m2/day CIVI x 2 days, every two weeks. Treatment will be performed on the scheduled day ± 7 days. In case of discontinuation of FOLFOX due to cumulative toxicity and administration as a single agent during the study, regorafenib for patient convenience will be administered 160 mg daily for 3 weeks on/1 week off. The 3 weeks on/1 week off schedule is supported by the single agent regorafenib data in colon cancer and GIST.
  Interventions: Drug: Regorafenib; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Regorafenib
  Other Names: (Bay 73-4506)
Drug: 5-Fluorouracil
Drug: Leucovorin
Drug: Oxaliplatin

SUMMARY:
The purpose of this study is to evaluate the effects, good and/or bad, of the drug regorafenib with chemotherapy regime (FOLFOX). This is a a Phase II trial that will study if this new treatment is effective and safe in patients with esophagus and stomach cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed metastatic or unresectable esophageal, gastroesophageal junction or gastric adenocarcinoma.
* Patient must have disease that can be evaluated radiographically. This may be measurable disease or non-measurable disease. Minimum indicator lesion size = 10 mm by helical CT or = 20 mm by conventional techniques. Pathological nodes must be = 15 mm by the short axis to be considered measurable.
* Subject must be able to swallow and retain oral medication
* Age 18 years or older.
* Karnofsky performance status > or = to 70%
* Peripheral neuropathy ≤ grade 1
* Hematologic (minimal values) White blood cell count > or = to 3000/mm3© Absolute neutrophil count > 1500 cells/ mm3 Hemoglobin > or = to 8.0 g/dl Platelet count > or = to 90,000 / mm3 Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphatase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer). Patients with alkaline phosphatase elevation secondary to the bony metastases rather than liver dysfunction may proceed with treatment on protocol after discussion with the principal investigator.
* Serum creatinine ≤ 1.5 x the ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test..
* Patients with prior deep vein thrombosis (DVT) or pulmonary embolism (PE) currently on an stable anticoagulation regimen with low molecular weight heparin (LMWH) or rivaroxaban will be permitted.

Exclusion Criteria:

* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:
* Congestive heart failure - New York Heart Association (NYHA) > Class II.
* Active coronary artery disease.
* Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
* Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE version 4.0 Grade 3 within 4 weeks prior to start of study medication.
* Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study.
* Active hepatitis B infection, active hepatitis C infection or known HIV carrier.
* Patient may not have received prior chemotherapy for metastatic or unresectable disease.
* Patients may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if more than 6 months have elapsed between the end of adjuvant therapy and registration.
* Patient may not have received prior 5-Fluorouracil, Leucovorin, Oxaliplatin or regorafenib. Patient may have received prior radiosensitizing doses of 5Fu if more than 6 months have elapsed between the end of adjuvant therapy and registration.
* Patient may not have had major surgical procedure within 4 weeks of registration.
* Patient may not have had radiation within 2 weeks of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FOLFOX Plus Regorafenib
Started | 39
Completed | 36
Not Completed | 3
Not completed — Not Eligible | 3

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOX Plus Regorafenib
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 58 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFOX Plus Regorafenib
Number analyzed (Participants) | 39
percentage of participants | 53 [38 to 71]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival will be measured from the start of treatment to death or last follow-up and will be estimated using the Kaplan-Meier method
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX Plus Regorafenib
Number analyzed (Participants) | 39
months | 14.2 [8.1 to 20.7]

3. Secondary Outcome: Overall Response Rate
Description: This is defined as the percentage of patients who have achieved either an objective complete or partial target lesion response that is confirmed on the RECIST 1.1 criteria. Complete or partial responses will be confirmed with repeat CT evaluation after 4 weeks.
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants with CR or PR
Arm/Group | FOLFOX Plus Regorafenib
Number analyzed (Participants) | 39
percentage of participants with CR or PR | 54 [37 to 70]

4. Secondary Outcome: Participants Evaluated for Toxicity
Description: Adverse events will be determined as per the NCI Common Toxicity Criteria, version 4.0. Toxicity during cycle 1 and subsequent cycles will be reported.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOX Plus Regorafenib
Number analyzed (Participants) | 39
Participants | 39

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | FOLFOX Plus Regorafenib
All-Cause Mortality (participants affected / at risk) | 30/39
Serious Adverse Events (participants affected / at risk) | 17/39
Other Adverse Events (participants affected / at risk) | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX Plus Regorafenib (N=39)
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Aspartate aminotransferase increased (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Blood bilirubin increased (Investigations) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 4
Gastrointestinal disorders -Other, specify (Gastrointestinal disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lipase increased (Investigations) | 1
Muscle weakness left-sided (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Serum amylase increased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 2
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 2
Thromboembolic event (Vascular disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Weight loss (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX Plus Regorafenib (N=39)
Fatigue (General disorders) | 31
Anemia (Blood and lymphatic system disorders) | 28
White blood cell decreased (Investigations) | 28
Peripheral sensory neuropathy (Nervous system disorders) | 27
Platelet count decreased (Investigations) | 27
Hypertension (Vascular disorders) | 25
Nausea (Gastrointestinal disorders) | 23
Neutrophil count decreased (Investigations) | 23
Alanine aminotransferase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 20
Mucositis oral (Gastrointestinal disorders) | 14
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 14
Alkaline phosphatase increased (Investigations) | 13
Anorexia (Metabolism and nutrition disorders) | 12
Diarrhea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 11
Vomiting (Gastrointestinal disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 9
Weight loss (Investigations) | 9
Blood bilirubin increased (Investigations) | 8
Hyponatremia (Metabolism and nutrition disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Edema limbs (General disorders) | 4
Lymphocyte count decreased (Investigations) | 4
Paresthesia (Nervous system disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Fever (General disorders) | 3
Headache (Nervous system disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
INR increased (Investigations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Small intestinal mucositis (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT01913639/Prot_SAP_000.pdf